CLINICAL TRIAL: NCT06382909
Title: Effects of the Probiotic k11-tmax on Symptoms and Inflammatory Markers in Children With Autism Spectrum Disorder
Brief Title: Effect of Probiotic Compound K11T e K11TMax in ASD
Acronym: ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deivis de Oliveira guimaraes (Network)
Collaborators: SENAI CIMATEC (Other)
Responsible Party: Sponsor-Investigator, Deivis de Oliveira guimaraes, Director of Research, Gon1 Gestao de Projetos
Organization: Gon1 Gestao de Projetos (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202302
Record Dates: First submitted 2024-03-28; First posted 2024-04-24 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Autism Spectrum Disorder
Keywords: intestinal inflammatory; cognitive; probiotics; asd; Gut Microbiota; Biomarkers
MeSH Terms: conditions — Autism Spectrum Disorder; Child Development Disorders, Pervasive | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, with placebo control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mix Probiotic K11T with out vitamins (Active Comparator): Drug-1: K11T
  1 dose/day Orally
  Interventions: Dietary Supplement: Inflammatory level; Dietary Supplement: Cognitive assessment; Dietary Supplement: Pedagogical assessment
- Mix Probiotic K11TMAX with vitamins (Active Comparator): Drug-1: K11Tmax
  1 dose/day Orally
  Interventions: Dietary Supplement: Inflammatory level; Dietary Supplement: Cognitive assessment; Dietary Supplement: Pedagogical assessment
- Placebo drugs (Placebo Comparator): Placebo
  1 dose/day Orally
  Interventions: Dietary Supplement: Inflammatory level; Dietary Supplement: Cognitive assessment; Dietary Supplement: Pedagogical assessment

INTERVENTIONS:
Dietary Supplement: Inflammatory level — Quantification of C-reactive Protein (PCR) Quantification of serum cortisol Insulin quantification Prolactin quantification Fecal calprotectin dosage
Dietary Supplement: Cognitive assessment — Neurological assessment Psychiatric assessment
Dietary Supplement: Pedagogical assessment — Sociopedagogical assessment

SUMMARY:
The research is characterized as a randomized, double-blind clinical trial (phase III) in which administered the probiotic K11-T (with and without added amino acids, fatty acids and vitamins) to children between 3 and 11 years old with Autism Spectrum Disorder - ASD, being subsequently assessed outcomes related to inflammatory markers and neuropsychiatric and sociopedagogical criteria. To this end, the study will create three groups, one of which will be a control group, which will receive a placebo, the other will receive the probiotic without micronutrients and another will receive the probiotic with added nutrients.

DETAILED DESCRIPTION:
To evaluate the effectiveness of probiotic compounds K11-T and K11-Tmax (enriched with amino acids, acids fatty acids and vitamins), in its solid and nano-encapsulated formulation to improve the criteria neuropsychiatric, sociopedagogical and inflammatory disorders in children with ASD.

Secondary:

* Characterize the sample of individuals with ASD who will participate in the study through a questionnaire with sociodemographic and pedagogical data such as: Age in years; gender in percentage terms of the sample according to female or male; Weight in kg; Height in centimeters; Time since diagnosis of ASD in years and presence of psychiatric or neurological comorbidities in percentage terms of the sample.
* Investigate the association between probiotic consumption and neuropsychological results using the scale unit validated in the literature Vineland Adaptive Behavior Scales - Third Edition (Vineland-3) in the questionnaire format answered by parents/guardians of the child with ASD;
* Investigate the association between probiotic consumption and the change of psychiatric parameters through the application of the validated Autism Diagnostic Observation Schedule (ADOS) scale with children with ASD,
* Investigate the association between probiotic consumption and the change of psychopedagogical parameters using the Childhood Autism Rating Scale (CARS) validated in the literature, which will be answered by the teachers responsible for each child participating in the study;
* Analyze the possible effect of probiotics on inflammatory aspects in individuals with ASD, through serum (Insulin, C-Reactive Protein, Prolactin and Cortisol) and fecal (fecal calprotectin) biomarkers;
* Analyze the difference of using the K11-Tmax version, enriched with supplements, on the neuropsychological, psychiatric and psychopedagogical outcomes described above in comparison to the group that used K11-Tmax alone.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must have a confirmed diagnosis of ASD carried out by qualified professionals, in accordance with the criteria established in the Diagnostic Manual and Statistics of Mental Disorders (DSM-5) or other diagnostic classification recognized.
* The study will include children and adolescents in the specific age range of 3 to 11years.
* Be regularly enrolled in a public or private school, or in a learning center special education.
* Absence of decompensated clinical or psychiatric comorbidities;
* Informed consent: Legal guardians must provide a informed consent, understanding the study objectives, procedures involved, the risks and benefits, as well as the freedom to withdraw from the study at any time. anytime.
* Informed Assent: Children ages 7 to 11 must provide an informed consent, understanding the objectives of the study, the procedures involved, the risks and benefits, as well as the freedom to withdraw from the study at any time. anytime.

Exclusion Criteria:

* - Concomitant restrictive medical conditions that may interfere with the results of the study, such as serious gastrointestinal diseases, significant metabolic diseases or immunodeficiencies.
* Use of specific medications such as broad-spectrum antibiotics or immunosuppressive medications during the follow-up period.
* Allergies or intolerances to components of the probiotics that will be administered.
* Previous or current participation in recent clinical studies with interventions different therapies.
* Uncontrolled heart conditions or serious unstable medical illnesses.
* Impossibility of being present on the pre-determined assessment dates clinics.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 505 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
Inflammation biomarker 1 | 90 days (Day 0, Day 45 and Day 90)
  Quantify inflammatory markers through blood collection:
  Quantification of C-reactive Protein (CRP) - results in mg/dL
Inflammation biomarker 2 | 90 days (Day 0, Day 45 and Day 90)
  Quantify inflammatory markers through blood collection: Serum Cortisol Quantification - results will be expressed in mcg/dL;
Inflammation biomarker 3 | 90 days (Day 0, Day 45 and Day 90)
  Quantify inflammatory markers through blood collection: Insulin Quantification - the results will be expressed in mcUI/ml;
Inflammation biomarker 4 | 90 days (Day 0, Day 45 and Day 90)
  Quantify inflammatory markers through blood collection: Prolactin Quantification - results will be expressed in ng/dL
Inflammation biomarker 5 | 90 days (Day 0, Day 45 and Day 90)
  Quantify inflammatory markers through blood collection: Fecal Calprotectin Measurement - expressed in μg/g
Neuropsychological Assessment | 90 days (Day 0, Day 45 and Day 90)
  involves a multidisciplinary approach, considering different aspects of neuropsychological functioning. Standardized analysis will be conducted using the Vineland Adaptive Behavior Scales - Vineland-3. The forms will be completed in their self-administered version by parents/caregivers and teachers, under the supervision of a qualified and trained health professional. Vineland-3 assesses adaptive behavior by dividing it into five domains: communication skills, daily living skills, socialization skills, motor skills and maladaptive/behavioral skills of the child. Those responsible will respond to the items in each domain on a scale ranging from 0 to 2, with 0 being never; 1 sometimes and 2 often. To calculate the final score, the scores are transformed into a population average of 100 based on age and a standard deviation of 15 according to the specific and standardized manual for the scale. A higher score indicates greater adaptive functioning.

SECONDARY OUTCOMES:
Psychiatric Assessment | 90 days (Day 0, Day 45 and Day 90)
  The ADOS-2 (Autism Diagnostic Observation Schedule, Second Edition) observational assessment will be applied. This is a standardized assessment that involves direct observation of the child in different situations and social interactions. The evaluated parameters are divided into 5 items according to the psychiatric criteria for ASD diagnoses by the Diagnostic and Statistical Manual of Mental Disorders (DSM): language and communication; reciprocal social interaction; play and imagination; stereotypical behaviors and restricted interests and, finally, atypical behaviors. The observation lasts 60 minutes and will be carried out by trained and qualified professionals supervised by a reference neuropsychologist. After applying the ADOS, the domains are coded on a scale that varies from 0 to 3 points, where 0 indicates that the child has a certain ability and 3 indicates abnormal or dysfunctional behavior.
Psychopedagogical Assessment | 90 days (Day 0, Day 45 and Day 90)
  Will be carried out using a questionnaire validated in literature in the version translated into Portuguese, called the Childhood Autism Rating Scale (CARS). It consists of a scale with fifteen parameters on the symptoms of autism spectrum disorder in children, which include: interpersonal relationships, imitation, emotional response, body use, use of objects, response to changes, visual response, auditory response, response and use of taste, smell and touch, fear or nervousness, verbal communication, non-verbal communication, level of activity, level and consistency of intellectual response and finally a general parameter of that individual's autism. Variations from 1 to 4, with number 1 corresponding to no difficulty in performing that skill until 4 being severe difficulty. If you are between 15 and 30 years old, you do not have autism; 30 to 36 mild to moderate autism and 36 to 60 correspond to severe autism.

OTHER OUTCOMES:
Comparative of outcomes between arm that took K11-T and arm that took K11-Tmax. | 90 days (Day 0, Day 45 and Day 90)
  Comparative of all outcomes from arm k11-T and K11-Tmax. Results will be expressed in %.

CONTACTS AND LOCATIONS:
Overall Officials: Deivis O Guimaraes, PhD student, Study Director — GON1 P&D
Locations (2):
- Brazil (2):
  - Gon1 gestora de Projetos, Vitória, Espírito Santo
  - Gon1 P&D, Vitória, Espírito Santo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: International Contract Research Organization — http://www.gon1.com.br
- See also: Ethics and research committee — http://www.uvv.br

DOCUMENTS (2):
  • Study Protocol (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT06382909/Prot_000.pdf
  • Informed Consent Form (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT06382909/ICF_001.pdf